CLINICAL TRIAL: NCT01894633
Title: Phase II Randomized, Double Blind, Placebo Controlled Study of Whole-brain Irradiation With Concomitant Daily-dose Chloroquine for Brain Metastases.
Brief Title: Study of Whole-brain Irradiation With Chloroquine for Brain Metastases
Acronym: CLQ
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, Principal Investigator, Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CD-449-08
Record Dates: First submitted 2013-06-29; First posted 2013-07-10 (Estimated); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Brain Metastasis
Keywords: Prophylactic Cranial Irradiation; Metastasis; Cloroquine
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis | interventions — Chloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chloroquine, radiosensitizer (Experimental): The patients in the Chloroquine group received 30 Gy of total brain radiotherapy in 10 daily fractions from Monday to Friday. Furthermore, the CLQ plus WBI arm received a daily single dose of 150 mg CLQ po 1 hour prior to the radiation treatment, beginning during the first radiotherapy fraction and continuing for 28 days.
  Interventions: Drug: Chloroquine; Radiation: Total brain radiotherapy
- Placebo (Placebo Comparator): 30 Gy of whole-brain radiotherapy in 10 daily fractions and an oral matching placebo for 28 days
  Interventions: Radiation: Total brain radiotherapy

INTERVENTIONS:
Drug: Chloroquine — The patients in the Chloroquine group received 30 Gy of total brain radiotherapy in 10 daily fractions from Monday to Friday. Furthermore, the Chloroquine plus WBI arm received a daily single dose of 150 mg CLQ po 1 hour prior to the radiation treatment, beginning during the first radiotherapy fraction and continuing for 28 days
  Other Names: Aralen
  Arms: Chloroquine, radiosensitizer
Radiation: Total brain radiotherapy — 30 Gy in 10 daily fractions from Monday to Friday

SUMMARY:
Background and purposes:Chloroquine (CLQ), an antimalarial drug, has a lysosomatrophic effect associate with increase the sensibility of Radiation through leakage of hidroliticenzimes, increase of apoptosis, autophagy mediated by lysosomalhidrolases and increase of oxidative stress "in vitro". In this phase II study we evaluated the efficacy and safety as radiosensitizing of the Chloroquine plus concomitant 30 Gray (Gy) of Whole-brain irradiation (WBI)in patients with brain metastases (BM) from solid tumors.

DETAILED DESCRIPTION:
Seventy-three eligible patients were randomized. Thirty-nine patients received WBI (30 Gy in 10 fractions over 2 weeks) concomitant with 150 mg of CLQ for 4 weeks (the CLQ group). Thirty-four patients received the same schedule of WBI concomitant with a placebo for 4 weeks (the control arm). All the patients were evaluated for quality of life (QoL) using the EORTC QLQ-C30 questionnaire (Mexican version) before beginning radiotherapy and one month later.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age
* At leat one brain metastasis MRI
* KPS 70 or more
* RTOG-RPA I or II
* Basic Laboratory requirements

Exclusion Criteria:

* Candidates for radiosurgery, neurosurgery
* Patients treated with radiotherapy before entered to the study

Ages: 46 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2011-05; Primary Completion 2012-04 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Every third month after randomization until 24 months follow-up. Measured by brain MRI
  Corresponding Complete plus Partial Response according with RECIST 1.1 Criteria

SECONDARY OUTCOMES:
Central Nervous System Progression Free Survival | From time to progression to 24 months follow up
  Clinical o radiological brain progression or death. Radiological Progression is measured by RECIST 1.1 Criteria

OTHER OUTCOMES:
Quality of life in brain metastases | The quality of life questionnaires were completed 1 day before radiotherapy began and 1 month later.
  The 30-item EORTC Quality of Life (QoL) Questionnaire (EORTC QLQ-C30) version 3.0 (Mexican version) was used in this trial. The EORTC QLQ-C30 v3 consisted of five multi-item functional scales, three symptom scales, a global health status/QoL scale, and six single items

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Arrieta, MD, Principal Investigator — Instituto Nacional de Cancerologia, Columbia
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Mexico City, Mexico